CLINICAL TRIAL: NCT06519240
Title: A Prospective Blinded Pilot Study Evaluating the Sensitivity and Specificity of 18F Fluorodeoxyglucose PET CT Imaging (a Non-invasive Imaging Tool) for the Diagnosis of Rejection in Heart Transplant Recipients.
Brief Title: A Pilot Study Evaluating the Potential of 18F Fluorodeoxyglucose PET-CT Imaging in Diagnosing Cardiac Rejection.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 335590/1660859/37/429
Record Dates: First submitted 2024-05-02; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Transplant Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with a diagnosis of cardiac rejection (Active Comparator): Based on heart muscle biopsy findings. Subjects must have no significant coronary disease within the last 12 months (with a confirmatory angiogram, computed tomography coronary angiogram, myocardial perfusion scan, cardiac magnetic resonance imagining, or other coronary ischaemia test.
  Interventions: Radiation: 18F-Fluorodeoxyglucose Positron Emission Tomography-computed Tomography (18F-FDG PET CT)
- Patients with no evidence of cardiac rejection (Active Comparator): Based on heart muscle biopsy findings
  Interventions: Radiation: 18F-Fluorodeoxyglucose Positron Emission Tomography-computed Tomography (18F-FDG PET CT)

INTERVENTIONS:
Radiation: 18F-Fluorodeoxyglucose Positron Emission Tomography-computed Tomography (18F-FDG PET CT) — Each participant will prepare for their study PET CT by following an initial 18 hour of zero carbohydrate diet followed by another 18 hours of fasting (water allowed). After confirming preparation, each study participant will have a single rest rubidium and 18F-FDG PET CT scan.

SUMMARY:
This pilot study aims to assess whether 18F-FDG PET CT imaging has the potential in diagnosing cardiac rejection. The investigators aim to recruit 20 heart transplant subjects within two groups of 10 subjects each. One group will have participants with definite rejection and the other group will have participants with definite no rejection. Subjects will be placed into study groups based on their heart muscle biopsy, echocardiogram, clinical symptoms, ECG, and presence or absence of donor specific antibodies. Each group will then undertake a 18F-FDG PET CT scan to identify whether this imaging modality has a role in identifying cardiac rejection. The study subjects and the research team will be blinded to the results of the PET CT until the end of the study.

DETAILED DESCRIPTION:
Approximately 12% of heart transplant recipients are treated for cardiac rejection during their first year of follow-up. Rejection is the cause of death in 8-10% of cases in the first three years. Currently, to diagnose cardiac rejection, patients require radiological imaging (for example echocardiography, or cardiac magnetic resonance imaging), and histological sampling, obtained invasively by performing a heart muscle biopsy ("endomyocardial biopsy").Biopsy is an invasive procedure with a serious risk of complications including cardiac tamponade and death. In addition, there are issues relating to sampling errors, as well as the interpretation of results, which can be semi-objective and challenging. Furthermore, as it is an invasive procedure, having a biopsy can cause anxiety and discomfort for patients. There is a clear need for a technique to diagnose cardiac rejection non-invasively, which can yield reliable and accurate results, permitting the prompt commencement of treatment.

Some studies in animals, and preliminary studies in humans, have shown potential for '18F-FDG PET CT' imaging to tackle this problem in diagnosing cardiac rejection. There is a clear need to undertake a large study, but it is not clear at this preliminary stage if this is feasible.

The investigators aim to perform this pilot study to determine if 18F-FDG PET CT imaging is acceptable for heart transplant patients, and to assess if it has the potential to diagnose cardiac rejection when compared to endometrial biopsy. It will also help provide data to assess sample size requirements to undertake a larger diagnostic study in the future. If this imaging modality is found to be beneficial, cardiac rejection may be reliably diagnosed sooner, resulting in prompt treatment and improvement in quality of life, with better prognosis in heart transplant recipients.

Each group, would undertake a resting Rubidium PET scan, jointly with a FDG PET scan at the same visit to exclude cardiac injury from previous cardiac events, and to assess heart function. An experienced consultant in nuclear medicine (who will remain blinded to the patient identification and medical history) will report the findings of the imaging to the study investigators.

ELIGIBILITY:
Inclusion Criteria:

* All heart transplant recipients with definite cardiac rejection or definite no rejection with evidence of no significant coronary disease within the last 12 months (e.g with any of the following tests (1)angiogram (2) CTCA (3) MPS (4) CMR (5) other coronary ischaemia test)

Exclusion Criteria:

* Unable to have a PET CT scan or comply with the dietary protocol
* Age less than 18 years old
* Unable to consent
* Presence of significant coronary disease or coronary ischaemia
* Insulin dependent diabetics
* Pregnant or breast feeding individuals

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-10-02 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Define the sensitivity and specificity of FDG PET CT in the diagnosis of cardiac rejection, when compared to the current clinical standard (cardiac biopsy and Echocardiography) | 18 months
  We aim to confirm the sensitivity and specificity of FDG PET CT in diagnosing cardiac rejection

SECONDARY OUTCOMES:
Practicality and acceptability of FDG PET CT imaging to patients | 18 months
  The investigators will aim to undertake a patient survey within 48 hours of the study taking place to ascertain the subjects whether undertaking FDG-PET CT imaging to patients is practical and acceptable to patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mansimran Dulay, MBBS MRCP, Study Director — Royal Brompton and Harefield Hospital

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD)

REFERENCES:
- [Result] Daly KP, Dearling JL, Seto T, Dunning P, Fahey F, Packard AB, Briscoe DM. Use of [18F]FDG Positron Emission Tomography to Monitor the Development of Cardiac Allograft Rejection. Transplantation. 2015 Sep;99(9):e132-9. doi: 10.1097/TP.0000000000000618. PMID 25675207